CLINICAL TRIAL: NCT03384030
Title: Exploration of the Modulation of Skin Microbiota and Odor Components by Introduction of Stress in Healthy Male Subjects
Acronym: MOIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL62290.041.17
Record Dates: First submitted 2017-11-07; First posted 2017-12-27 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2017-12

CONDITIONS: Emotional Stress
Keywords: Malodor; Stress; STMST
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention. 30 healthy males are subjected to the adapted STMST to induce emotional sweating.
Masking Description: Subjects will be kept naïve with respect to the fact that stress responses are the primary responses of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adapted STMST (Experimental): Participants are subjected to the adapted STMST to induce emotional sweating.
  Interventions: Other: adapted STMST

INTERVENTIONS:
Other: adapted STMST — Participants are subjected to the adapted STMST to induce emotional sweating.

SUMMARY:
In the MOIST study it will be assessed whether the adapted Sternberg short-term working memory task (STMST) is an effective method to induce malodor formation by emotional stress, as assessed by expert assessments of stress-induced malodor formation in the armpits of 30 healthy male volunteers.

Before, during and after being exposed to the adapted version of the STMST, saliva will be collected to determine cortisol levels, subjects have to rate their momentary feelings of anxiety and embarrassment and heart rate variability will be monitored continuously with a wireless signal transmission device. Before and after exposure to the adapted STMST, malodor levels will be assessed by two expert judges, axillary volatiles will be collected by cup scrubbing and microbiota samples will be taken to determine microbial species.

DETAILED DESCRIPTION:
Stress is a primary physiological response to physical and/or social threats resulting from a complex interplay of neurophysiological and psychological factors. Cognitive interpretations of social-evaluative threats have been found to be very potent emotional stressors. Apocrine sweat glands are stimulated by emotional stress, fear or mental tension. Upon secretion, apocrine sweat is odorless. By enzymatic action of the bacterial microbiome on apocrine sweat in particular, body malodor is formed. This is perceived as offensive by most societies. As a result, self-confidence and social relationships can be influenced by undesired body odor. A good understanding of the complex sweat-microbiome interactions leading to malodor formation is required for the development of effective malodor remedies.

In the MOIST study it will be assessed whether the adapted Sternberg short-term working memory task (STMST) is an effective method to induce malodor formation by emotional stress, as assessed by expert assessments of stress-induced malodor formation in the armpits of 30 healthy male volunteers.

Before, during and after being exposed to the adapted version of the STMST, saliva will be collected to determine cortisol levels, subjects have to rate their momentary feelings of anxiety and embarrassment and heart rate variability will be monitored continuously with a wireless signal transmission device. Before and after exposure to the adapted STMST, malodor levels will be assessed by two expert judges, axillary volatiles will be collected by cup scrubbing and microbiota samples will be taken to determine microbial species.

ELIGIBILITY:
Inclusion Criteria:

1. Male;
2. Age 18-34 yrs;
3. BMI between 18,5-25 kg/m2;
4. Healthy as assessed by the NIZO lifestyle and health questionnaire;
5. Non-smoking;
6. Signed informed consent;
7. Malodor score ≥ 4≤ 8 as assessed by malodor judges
8. Access to internet;
9. Voluntary participation;
10. Willing to accept disclosure of the financial benefit of participation in the study to the authorities concerned;
11. Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for the study for at least 15 years;
12. Willing to accept information-transfer concerning participation in the study, or information regarding health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner;
13. Willing to comply with study procedures.

Exclusion Criteria:

1. Alcohol consumption > 15 units/week and > 3/day;
2. Drug abuse;
3. Former participation in a cognitively challenging computer task or mental performance test;
4. Heavy exercise or sports training > 10 hours/week;
5. Hyperhidrosis , Hypohidrosis or Anhidrosis;
6. Known allergy to cosmetics;
7. Mental status that is incompatible with the proper conduct of the study;
8. Participation in any scientific study with oral, intravenous or inhalatory administration of any substances during two (2) months before study start that could interfere with the MOIST study;
9. Psychiatric disorders;
10. Use of anti-anxiety medications or beta-blockers, statins or blood pressure medication;
11. Use of antibiotics during the six (6) months prior to study start;
12. Use of topical medications in underarm area during 2 weeks prior to study start;
13. Recurring infections, boils, abscesses or lymph node enlargement in the underarm and ;
14. Active eczema or psoriasis on any portion of the body.
15. Personnel of the research institute(s) involved in execution of the study, their partner and their first and second degree relatives;
16. Not having a general practitioner, not allowing disclosure of participation to the general practitioner or not allow to inform the general practitioner about abnormal results.

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity is self-reported by the subjects through a questionnaire.
Enrollment: 30 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-03-17 (Actual)

PRIMARY OUTCOMES:
stress-induced malodor formation | Change from baseline malodour formation 20 min, 40 min, and 60 minutes after the start of exposure to the adapted STMST
  Expert assessments of stress-induced malodor formation by emotional stress in the armpits of healthy male volunteers

SECONDARY OUTCOMES:
Salivary cortisol | Change from baseline salivary cortisol 5 min, 20 min, 30 min, 40 min, 50 min, 60 min, and 70 minutes after the start of exposure to the adapted STMST
  Emotional stress in healthy male volunteers as assessed by cortisol in saliva
Self-assessed mood state | Change from baseline self-assessed mood state 5 min, 20 min, 30 min, 40 min, 50 min, 60 min, 70 min, and 90 minutes after the start of exposure to the adapted STMST
  Emotional stress in healthy male volunteers as assessed by self-assessed mood state (VAS)
Malodor compounds formation | Change from baseline malodour compounds formation 75 minutes after the start of exposure to the adapted STMST
  The malodor compounds formation as assessed by GC-MS/MS analyses during conditions of emotional sweating

CONTACTS AND LOCATIONS:
Overall Officials: Melle van Schaik, Study Director — NIZO Food Research
Locations (1):
- NIZO, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No